CLINICAL TRIAL: NCT03244072
Title: Safety and Efficacy of Intracameral Zimoxin (0.1% Moxifloxacin Solution) for Prevention of Endophthalmitis After Cataract Surgery
Brief Title: Safety and Efficacy of Intracameral Zimoxin for Prevention of Endophthalmitis After Cataract Surgery
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jason Ahee, M.D. (Industry)
Responsible Party: Sponsor-Investigator, Jason Ahee, M.D., Medical Director, Zion Therapeutics, LLC
Organization: Zion Therapeutics, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PIND 134134
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Endophthalmitis
MeSH Terms: conditions — Endophthalmitis | interventions — Moxifloxacin; Exercise; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): Intracameral injection of moxifloxacin solution after cataract surgery
  Interventions: Drug: Moxifloxacin
- Placebo group (Placebo Comparator): Intracameral injection of placebo after cataract surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxifloxacin — Intracameral injection
  Other Names: active
  Arms: Treatment group
Drug: Placebo — intracameral injection
  Other Names: sham
  Arms: Placebo group

SUMMARY:
Intracameral injection of 0.1% moxifloxacin solution after cataract surgery to prevent endophthalmitis

DETAILED DESCRIPTION:
Subjects will receive either intracameral injection of 0.1% moxifloxacin solution or placebo after cataract surgery. They will be followed for one month to determine if there is a statistically significant difference in the incidence of endophthalmitis.

ELIGIBILITY:
Inclusion Criteria:

* visually significant cataracts

Exclusion Criteria:

* allergy to fluoroquinolones, cobalamin (B12)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60000 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Endophthalmitis after cataract surgery | Subjects will undergo eye examinations at one day, one week, and one month post-operatively
  Subjects will be followed after cataract surgery and have post-operative eye examinations to determine if infection in the eye (endophthalmitis) occurs during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Ahee, M.D., Principal Investigator — Zion Therapeutics, LLC
Locations (1):
- Zion Eye Institute, St. George, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided